CLINICAL TRIAL: NCT06937463
Title: Feasibility of Virtual Reality-Based Rehabilitation in Patients With Limited Mobility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: UNIST (Ulsan National Institute of Science and Technology) (Unknown)
Responsible Party: Principal Investigator, Won Kim, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2024-1735-0010
Record Dates: First submitted 2025-04-20; First posted 2025-04-22 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Bed-ridden Patient
Keywords: bed-ridden patients; Motion recognition
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- This is a study on the recovery of physical function in bed patients through a digital rehabilitatio (Experimental): This is a study on the recovery of physical function in bed patients through a digital rehabilitation exercise system
  Interventions: Behavioral: Rehabilitation

INTERVENTIONS:
Behavioral: Rehabilitation — This is a study on the recovery of physical function in bed patients through a digital rehabilitation exercise system

SUMMARY:
Study title:

Customized Evidence-Based Motion Recognition Rehabilitation Exercise System for Bed Stabilization Patients

the purpose of the study This study aims to evaluate the effectiveness of rehabilitation programs using motion recognition-based games for patients who are bedridden in hospital settings. The main purpose of the study is to determine whether digital rehabilitation can substantially contribute to the improvement and recovery of physical function in patients with limited physical functioning.

a study participant The study involved 28 adult patients who were hospitalized while lying in bed at a hospital. Participants use Nintendo Ring Fit, which provides a motion-aware-based game rehabilitation exercise program, and a personalized exercise plan is provided for each patient's physical condition.

research methodology Exercise Protocol: Participants will perform a personalized exercise program for two weeks through Nintendo Ring Fit. The exercise lasts about 30 minutes, once a day and is supported by a therapist. Exercise intensity and type are adjusted to suit the patient's physical condition so that they proceed safely.

Monitoring safety and effectiveness: Keep track of participants' physical functions (e.g., strength, mobility, etc.) during the study, and constantly monitor for any inconveniences or side effects that may occur during exercise sessions. This closely checks patients' motor responses and ensures safety.

the duration of the study The study runs from September 2024 to December 2025, during which participants will undergo rehabilitation exercises using motion recognition-based games.

Estimated results The study is expected to demonstrate that digital rehabilitation programs can be a safe and effective treatment option for patients who are bedridden in hospital settings. In addition, the findings will contribute to improving in-hospital rehabilitation practices and promoting physical recovery.

Safety Considerations All exercises conducted in this study are designed with safety as the top priority, and exercise intensity is adjusted to low intensity. If patients experience discomfort or side effects during the exercise, they are monitored closely and allowed to take the necessary action immediately. All exercises are conducted safely under the supervision of a medical professional.

DETAILED DESCRIPTION:
Research Plan Summary 제목: Customized Evidence-Based Motion Recognition Rehabilitation Exercise System for Bed Stabilization Patients

Objective:

This study aims to evaluate the validity of the intervention by analyzing the effectiveness, safety, and compliance of the rehabilitation exercise program using Nintendo Ring Fit™ for patients with limited behavior.

Senior Investigator: Dr. Kim Won Co-investigators: Dr. Cha Seung-woo, Dr. Choi Jong-won, and Researcher Kim Se-eun Agency: Asan Medical Center, Seoul Study Participants: Patients with a functional outpatient category (FAC) score of 3 or less among hospitalized patients at Asan Medical Center in Seoul.

Study Design: A prospective cohort clinical study of 28 participants meeting inclusion and exclusion criteria.

Evaluation Method: Design a rehabilitation exercise program with possible movements while lying or sitting based on Exer-gaming (Nintendo Ring Fit™). At Asan Medical Center in Seoul, rehabilitation exercise intervention is performed for patients who meet the above conditions by applying the program in a way that is possible according to the individual functions of the patients. This intervention is conducted for a maximum of two weeks and is applied within 30 minutes per session.

1. background of study In addition to central nervous system injuries, many of the patients admitted to the tertiary hospital often have limited mobility due to Intensive Care Unit Acquired Weakness (ICU-AW), Sarcopenia, and general weakness due to various acute medical conditions. Although the survival rate has increased due to recent advances in medical technology, the prevalence of these conditions is also increasing (B. Jonghe, 2009).

   This behavioral limitation implies several risk factors for patients. It can act as an independent risk factor for medical complications such as poor quality of life of an individual, increased risk of falls, hospital-acquired pneumonia, urinary tract infections, etc. (X. Wu, 2018). Even after being discharged from the hospital, some patients may face difficulty recovering from pre-existing physical functions (R. Zorowitz, 2016).

   To address these issues, rehabilitation therapy is being actively studied in the clinical setting as a very important intervention method. For example, in a study by Morris PE et al. (2008), in ICU-AW patients **Early Mobilization**, which consists of a range from **passive range of motion** to **Active Transfer to Chair**, resulted in shorter ICU hospital stay and hospital stay, and shorter time to walk. In addition, the mortality and readmission rates within one year were lower than those of the control group.

   In a study by T. Sricharoenchai et al. (2014), as a result of performing early rehabilitation exercise intervention in a similar patient group, no side effects occurred enough to extend the hospitalization period, and it had a positive effect on the patients' function recovery. In addition, a study by Ogawa et al. (2021) reported that low-intensity muscle strength and aerobic exercise in patients with restriction of behavior diagnosed as Sarcopenia after cardiovascular surgery were effective in improving functions such as muscle mass and walking speed.

   These studies demonstrate that rehabilitation exercise therapy plays an important role in patients with limited behavior. However, most of the existing studies have been conducted in patients with central nervous system injuries or inpatient settings, and relatively few studies have been conducted on inpatients. In addition, most of the existing studies have limitations in that the intervention period is short, it is for patients living in the community who are not inpatients, or the function and performance evaluation is not quantitative.

   By supplementing these limitations, this study aims to evaluate the feasibility of a rehabilitation exercise program for inpatients with limited behavior using a commercialized Nintendo Ring Fit™ game. Through this, the effectiveness of exer-gaming rehabilitation exercise intervention is quantitatively measured, safety is reviewed, and compliance and satisfaction are evaluated to analyze the usefulness in the clinical field.
2. research objectives Develop rehabilitation programs and platforms for hospitalized patients and verify their feasibility and safety.
3. Estimated duration of study The study will run from the IRB approval date to July 31, 2026.
4. Study Participants and Methods 1) a study participant

Inclusion criteria:

* Patients with restricted mobility (FAC 3 or less) among those hospitalized for acute, surgical conditions

  * FAC 3: One guardian is required to supervise walking without physical contact
* A person who is 19 years of age or older and who has agreed to this study

Exclusion criteria:

-Those who are unable to cooperate in rehabilitation exercise programs due to inadequate levels of consciousness or cognition - those who have persistent biological instability

-A person who is unable to perform most of the exercise programs due to severe limitation of muscle strength or range of motion of the joint, disability of amputation, etc

* A person who needs to limit the movement required for the rehabilitation exercise program due to fracture or instability of the skeletal system- A person who is unable to cooperate with the rehabilitation exercise program due to poor vision or hearing
* Patients on mechanical ventilation for 24 hours

Target sample size and rationale:

This study is a pilot study, considering similar studies in the past, the above study period, and the environment of the hospital, the dropout rate of the patient group that can be secured during the study period is considered to be 28, and the possible patients are to be secured as subjects for the study.

2) a method of research Based on Exer-gaming (Nintendo Ring Fit™), we design a rehabilitation exercise program with possible movements while lying or sitting. At Asan Medical Center in Seoul, rehabilitation exercise intervention is conducted for patients who meet the above conditions by applying the program in a way that is possible according to the functions of each patient. This intervention is based on performing a total of 10 exercise interventions in a period of 2 weeks, but if it is not possible to perform it depending on the condition of the subject, it should be completed within 1 month. Apply within 30 minutes per session. Before the start of the intervention, the following items are investigated for the possibility of exercise motion. After that, during the intervention, whether the operation was implemented and the number of repetitions were investigated.

5. Statistical Analysis Principles and Methods

- Computational statistical processing is performed using SPSS and R programs, and the specific method is as follows, and the statistical significance level is set to p<0.05.- The patient's performance, severity, and assistance are described in a descriptive manner.- Chi-square test and logistic regression are used to analyze categorical dependent variables, and Wilcoxon signed rank test, Friedman test, and Spearman correlation are used to analyze continuous dependent variables (function before and after intervention, exercise performance level, patient report results, etc.).

6. criteria for withdrawal of participants

Participants can withdraw from the study at any time. Other withdrawal criteria include:

Participants or legal guardians request withdrawal Find that participants are no longer or suitable for the study The decision of the investigator or the ethics committee is inappropriate.

7. anticipated side effects Side effects such as temporary shortness of breath, tachycardia, blood pressure changes, falls, and deviations can occur. However, since this intervention involves low-intensity exercise, serious side effects are less likely to occur. The risk of falling is considered to be minimal compared to rehabilitation performed outside of bed.

8. Early Termination Criteria

The study may be terminated early under the following conditions:

Participant withdrawal Discovery that the participant is unsuitable for the study Investigator or ethics committee judgment that the study should be discontinued If the ethics committee or institution decides the trial should be halted.

9. Ethical Considerations This study will be conducted in compliance with ethical guidelines approved by the Institutional Review Board (IRB). Informed consent will be obtained from participants or legal guardians, ensuring they fully understand the purpose, procedures, and potential risks of the study. All personal data will be anonymized to protect privacy.

10. Measures for Protecting Participant Privacy All personal data will be kept confidential. Data will be anonymized and stored securely, with access limited to the principal investigator and co-investigators. Video data will be encrypted and shared only with collaborating institutions.

ELIGIBILITY:
* Patients with restricted mobility (FAC 3 or less) among those hospitalized for acute, surgical conditions

  * FAC 3: One guardian is required to supervise walking without physical contact
* A person who is 19 years of age or older and who has agreed to this study

Exclusion criteria:

* Those who are unable to cooperate in rehabilitation exercise programs due to inadequate levels of consciousness or cognition - those who have persistent biological instability
* A person who is unable to perform most of the exercise programs due to severe limitation of muscle strength or range of motion of the joint, disability of amputation, etc
* A person who needs to limit the movement required for the rehabilitation exercise program due to fracture or instability of the skeletal system- A person who is unable to cooperate with the rehabilitation exercise program due to poor vision or hearing
* Patients on mechanical ventilation for 24 hours

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility | From enrollment to end of two-week treatment
  Enter the actual exercise time and number of exercises for the total exercise time to record whether the patient complies with the rehabilitation program.

SECONDARY OUTCOMES:
Safety | From enrollment to the end of treatment at 2 weeks
  Monitoring the number of occurrences of adverse events such as pain, falls, dizziness, and any other negative reactions during the rehabilitation sessions.

OTHER OUTCOMES:
Medical Research Council Sum Score (MRC-SS) | From enrollment to the end of treatment at 2 weeks
  Summation score of muscle strength based on MRC scale. Unit of Measure: Sum score (0 to 60, where a higher score indicates better overall muscle strength.)
Functional Ambulatory Category (FAC) | From enrollment to the end of treatment at 2 weeks
  Measurement of the level of ambulation and assistance required. Unit of Measure: FAC score (0 to 5, where a higher score indicates greater walking independence.)
Hand Grip Strength Test | From enrollment to the end of treatment at 2 weeks
  Measurement of grip strength using a dynamometer. Unit of Measure: Force (kg) (A higher value indicates better grip strength.)
Knee Extensor Test | From enrollment to the end of treatment at 2 weeks
  Assessment of knee extensor strength using a dynamometer. Unit of Measure: Force (N or kg) (A higher value indicates stronger knee extensor muscles.)
10-meter Walk Test (10MWT) | From enrollment to the end of treatment at 2 weeks
  Assessment of walking speed and functional mobility over a 10-meter distance. Unit of Measure: Time (seconds) or speed (m/s) (For time: A lower value indicates faster walking ability. For speed: A higher value indicates better walking performance.)
Mini-Mental State Examination (MMSE) | From enrollment to the end of treatment at 2 weeks
  Cognitive function assessment using the MMSE tool. Unit of Measure: MMSE score (0 to 30, where a higher score indicates better cognitive function.)
EQ-5D Health-Related Quality of Life | From enrollment to the end of treatment at 2 weeks
  Assessment of patient-reported quality of life using the EQ-5D questionnaire, covering mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Unit of Measure: Utility score (0 to 1) and VAS score (0 to 100)
Satisfaction | From enrollment to the end of treatment at 2 weeks
  Assessment of patient satisfaction with the Nintendo Ring Fit and its use during rehabilitation exercises. Measurement Tool: Overall satisfaction, interest about health, Nintendo Ring Fit questions, exercise intensity questionnaire (5-point Likert scale) Unit of Measure: Satisfaction score (1 to 5, where a higher score indicates greater satisfaction.)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Songpa-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
All individual patient data (IPD) used in this study will be handled in compliance with domestic privacy protection laws and relevant regulations. The privacy of study participants will be strictly safeguarded, and their personal information will not be used for purposes other than the study. When sharing data, only de-identified data that has been approved by the researchers after adequate request will be provided, and privacy protection and security will be prioritized throughout the process.